CLINICAL TRIAL: NCT04900077
Title: Short Term Effect of Carriere® Motion™ Appliance on Pharyngeal Airway Dimensions: A Prospective Controlled Clinical Study
Brief Title: Effect of Carriere® Motion™ Appliance on Airway Dimensions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Slaha Aljohani, Assistant Professor & Consultant of Orthodontics, King Abdulaziz University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 022-01-19; 1532-165-1440 (Other Grant/Funding Number: King Abdulaziz University Research Grants)
Record Dates: First submitted 2021-05-05; First posted 2021-05-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Effect of Carriere® Motion™ Appliance on Pharyngeal Airway Dimensions; Effect of Carriere® Motion™ Appliance on Skeletal and Dental Measurements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- treatment group (Experimental): treated by Carriere® Motion™ Appliance
  Interventions: Device: Carriere® Motion™ Appliance
- control group (No Intervention): no treatment

INTERVENTIONS:
Device: Carriere® Motion™ Appliance — class II malocclusion corrector
  Arms: treatment group

SUMMARY:
Objectives: to evaluate the effect of treatment with Carriere® Motion™ Appliance on pharyngeal airway, skeletal and dental dimensions using lateral cephalometric radiographs and to compare these changes with a control group.

Materials and Methods: a prospective controlled clinical study on 17 patients treated at King Abdulaziz university dental hospital, Jeddah, Saudi Arabia with a mean age of 15.25 ± 2.49 years with class II molar relationship (treatment group). They were treated with Carriere® Motion™ Appliance and initial and post treatment lateral cephalograms were taken to assess the effect of the appliance on the pharyngeal airway dimensions, skeletal and dental measurements. A matched sample of 18 untreated patients (with a mean age of 14.44 ± 2.25 years) acted as a control group. Independent sample T-test and paired T-tests were conducted. The significance level was set at P< 0.05.

Results: when the cephalometric changes associated with the treatment by Carriere® Motion™ Appliance were compared to the changes in the untreated control group, no significant differences were found between the groups in regard to the pharyngeal airway and the skeletal dimensions. The only significant difference between the two groups was in the proclination and the protrusion of the lower incisors. The treatment group showed significantly increased lower incisors proclination and protrusion (L1 to mand plane°= 3.38±2.6, L1-Apo= 0.99±1.45) compared to the control group (L1 to mand plane°=0.49±2.81, L1-Apo=0.39±1.86) (P<0.05).

Conclusion: treatment with Carriere® Motion™ Appliance does not have a significant effect on pharyngeal airway and skeletal dimensions. However, it significantly increases the lower incisors proclination and protrusion.

ELIGIBILITY:
Inclusion Criteria:

* Class II molar relationship.
* Full set of teeth from 1st molar to 1st molar.
* Age: between 12 and 20 years.

Exclusion Criteria:

* Craniofacial deformities.
* Previous orthodontic treatment.
* History of respiratory illness.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
cephalometric pharyngeal airway changes (linear cephalometric measurements in mm) | For the treatment group: when class I molar relationship achieved. For the control group: not more than 18 months interval between the two lateral cephalograms.

SECONDARY OUTCOMES:
skeletal and dental cephalometric changes (linear and angular cephalometric measurements) | For the treatment group: when class I molar relationship achieved. For the control group: not more than 18 months interval between the two lateral cephalograms.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia